CLINICAL TRIAL: NCT02094807
Title: A Prospective Randomized Controlled Trial of Pain as Indication for Operative Treatment of Traumatic Rib Fractures.
Brief Title: Pain as Indication for Operative Treatment of Traumatic Rib Fractures
Acronym: potf
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow inclusion rate. Awaiting results from NCT02132416.
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Eva-Corina Caragounis, MD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hg481115; epn887-13 (Registry Identifier: Ethical approval committe)
Record Dates: First submitted 2014-03-18; First posted 2014-03-24 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Trauma; Rib Fractures; Surgery; Pain
Keywords: prospective study; surgical management; rib fractures; trauma
MeSH Terms: conditions — Wounds and Injuries; Rib Fractures; Pain | interventions — Anti-Inflammatory Agents, Non-Steroidal; Tramadol; Diclofenac; Naproxen; Analgesics, Opioid; Oxycodone; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conservative management (Other): Not operated. Thoracic epidural anesthesia will be used togeteher with paracetamol. If not sufficient opioids and NSAID will be added.
  Interventions: Drug: NSAID; Procedure: thoracic epidural anesthesia; Drug: opioids; Drug: paracetamol
- Operative management (Active Comparator): Operative fixation of rib fractures. Thoracic epidural anesthesia will be used togeteher with paracetamol. If not sufficient opioids and NSAID will be added.
  Interventions: Drug: NSAID; Procedure: thoracic epidural anesthesia; Drug: opioids; Drug: paracetamol; Procedure: operative fixation of rib fractures

INTERVENTIONS:
Drug: NSAID — Will be used if other drugs are not tolerated.
  Other Names: Tramadol; Voltaren; Naprosyn; Diclofenac
Procedure: thoracic epidural anesthesia — Continous epidural anesthesia will be introduced by specialists in Anesthesia and Intensive care.
Drug: opioids — During firs 24 hours i.v will be used. Then slow releas tabletts will be preferred.
  Other Names: Oxycotin; Oxynorm; Oxycodone; Morfin
Drug: paracetamol — 100mg x 4 i.v. during the first 24 hours. Then orally 100mg x 4.
  Other Names: Paracet; Alvedon; Panodil
Procedure: operative fixation of rib fractures — Fractures will be stabilized on the outside of of the ribs.
  Other Names: Matrix RIB Fixation Systems (De Puy Synthes)
  Arms: Operative management

SUMMARY:
The purpose of this prospective randomized controlled study is to determine whether acute and chronic pain in patients who suffer multiple traumatic rib fractures is decreased after surgical management as compared to conservative management.

DETAILED DESCRIPTION:
Patients meeting the inclusion criteria and giving their informed consent will be enrolled in this prospective randomized controlled study. In total 60 patients will be randomized to either surgical or conservative management of rib fractures. 3D reconstructions of computed tomography images of the Thorax done at admission to hospital will be used in order to evaluate injury according to Lung Injury Scale and Chest wall Injury Scale and for calculating radiological lung volumes and plan surgical procedure in the intervention group. Surgery will be performed as soon as possible after randomization. MatrixRIB® (DePuy Synthes) Fixation system is used for stabilizing rib fractures with plates and angular locked screws. Unless there is a medical indication or the patient has a chest tube pre-operatively, thoracotomy will be avoided. In cases where thoracotomy is done the patients will receive an anterior and posterior chest tube and wound drain with active suction. All patients, both in the intervention and in the control group will be offered thoracic epidural anaesthesia. Broad-spectrum antibiotic therapy iv is given as long as the patient has chest tubes. Thrombotic prophylaxis with LMWH is given until the patient is mobilized but for a minimum of 7 days. Patients will be followed-up 6 weeks, 6 months and 1 year post-operatively by surgeon and physiotherapist. A low-dosage computer tomography of the thorax will be done after 6 months in order to evaluate healing of the rib cage, possible non-union or dysfunction of osteosynthetic material and measure remaining lung volume. This examination will be compared to the initial computer tomography image done when the patient was admitted. At follow-ups complaints, possible late complications, usage of analgesia and return to work will be recorded. Evaluated instruments, EQ-5D-5L, VAS with Pain-O-Meter (POM) and Disability Rating Index (DRI) will be used to evaluate quality of life, pain and physical function. Range of motion in the thorax, thoracic spine and shoulders will be evaluated for every patient. Breathing movements will be measured by using a Respiratory movement measuring instrument (RMMI, ReMo Inc) and lung function tests will be performed in a standardized manner.

ELIGIBILITY:
Inclusion Criteria:

Adults ≥18 years of age with traumatic rib fractures that meet the following 2 criteria:

1. A minimum of 4 rib fractures
2. Pain that requires analgesia in the form of opioids in equivalent doses of > 25 mg iv morphine daily

Exclusion Criteria:

1. Concurrent spinal cord injuries with paralysis
2. Severe head injury where normal level of consciousness is not present
3. Severe neurological and musculoskeletal diseases that influence the function of the thoracic wall and lung volumes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Pain: VAS (1-10) | 1 year
  VAS (1-10)

SECONDARY OUTCOMES:
time spent in hospital | 6 weeks
  Length of stay
EQ-5D-5L | 1 year
  Quality of Life
DRI | 1 year
  Function and Activity

OTHER OUTCOMES:
The total cost | 1 year
  Adding time spent in hospital, on ICU or high-care unit and time before return to work

CONTACTS AND LOCATIONS:
Overall Officials: Hans Granhed, MD PhD, Study Director — Sahlgrenska University Hospital; Eva-Corina Caragounis, MD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden